CLINICAL TRIAL: NCT01782677
Title: Bilateral Surgical Resection of Carotid Bodies in Patients With Systolic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noblewell (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIM-B
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Systolic Heart Failure; Peripheral Chemoreceptor Hypersensitivity
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bilateral Surgical Resection of Carotid Bodies (Experimental): Patients undergoing Bilateral Surgical Resection of Carotid Bodies.
  Interventions: Procedure: Bilateral Surgical Resection of Carotid Bodies

INTERVENTIONS:
Procedure: Bilateral Surgical Resection of Carotid Bodies

SUMMARY:
The primary aim of the study is to determine safety, tolerability and feasibility of bilateral carotid body resection in patients with systolic heart failure and peripheral chemoreceptor hypersensitivity. The secondary aim is to assess potential efficacy of bilateral carotid body resection.

ELIGIBILITY:
Inclusion Criteria:

* History of heart failure class II-III according to NYHA within at least 6 months prior to inclusion
* Stable clinical state within at least 4 weeks prior to inclusion
* Subject >= 18 years old
* Left ventricular ejection fraction ≤ 45% evaluated by transthoracic echocardiography (Simpson's method)
* Carotid body present in computer cervical angiotomography
* History of exacerbated peripheral chemoreceptor sensitivity determined as >0.6L/min/%SpO2
* Able and willing to give written informed consent

Exclusion Criteria:

* Unstable angina pectoris, coronary attack, coronary revascularization, exacerbation of heart-failure requiring hospitalization, clinically significant infection, surgery under general anesthesia within 3 months prior to inclusion
* History of stroke, transient ischemic attack (TIA), or clinically significant chronic neurological disorder
* History of heart transplant
* Pregnancy or anticipation of pregnancy
* Hemodialysis or peritoneal dialysis patients
* Obstructive carotid atherosclerotic disease with >50% stenosis
* COPD stage III and IV according to GOLD 2007
* Unable to perform the spiroergometric assessment
* Any significant anomaly in additional investigation which may increase the risk of study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Peripheral chemosensitivity | 4 weeks
  Change from baseline in peripheral chemosensitivity measured as ventilatory response to hypoxia using transient inhalation of nitrogen at 4 weeks.
Muscle sympathetic nerve activity | 4 weeks
  Change from baseline in muscle sympathetic nerve activity at 4 weeks.

SECONDARY OUTCOMES:
Exercise tolerance | 4 weeks
  Change from baseline in exercise tolerance (peak oxygen consumption, slope relating minute ventilation to carbon dioxide production, oxygen uptake efficiency slope, time of exercise, 6-minute walking test distance, New York Heart Association Class) at 4 weeks.
Quality of life | 4 weeks
  Change from baseline in quality of life (Kansas City Cardiomyopathy Questionnaire, visual analog scale) at 4 weeks.
Serum concentration of NT-proBNP | 4 weeks
  Change from baseline in serum concentration of NT-proBNP at 4 weeks.
Barosensitivity | 4 weeks
  Change from baseline in barosensitivity at 4 weeks.
Peripheral chemosensitivity | 8 weeks
  Change from baseline in peripheral chemosensitivity measured as ventilatory response to hypoxia using transient inhalation of nitrogen at 8 weeks.
Muscle sympathetic nerve activity | 8 weeks
  Change from baseline in muscle sympathetic nerve activity at 8 weeks.
Exercise tolerance | 8 weeks
  Change from baseline in exercise tolerance (peak oxygen consumption, slope relating minute ventilation to carbon dioxide production, oxygen uptake efficiency slope, time of exercise, 6-minute walking test, New York Heart Association Class) at 8 weeks.
Sleep pattern in PSG | 8 weeks
  Change from baseline in sleep pattern in PSG (apnoea-hypopnoea index, percentage of central and obstructive episodes, average oxygen saturation, number of arousals, average duration of apnoeic and hypopnoeic episodes) at 8 weeks.
Quality of life | 8 weeks
  Change from baseline in quality of life (Kansas City Cardiomyopathy Questionnaire, visual analog scale) at 8 weeks.
Heart function and morphology | 8 weeks
  Change from baseline in heart function and morphology (transthoracic echocardiography) at 8 weeks.
Serum concentration of NT-proBNP | 8 weeks
  Change from baseline in serum concentration of NT-proBNP at 8 weeks.
Barosensitivity | 8 weeks
  Change from baseline in barosensitivity at 8 weeks.
Arrhythmia burden | 8 weeks
  Change from baseline in arrhythmia burden (24 hour ECG tape) at 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Ponikowski, Prof., Principal Investigator — 4. Wojskowy Szpital Kliniczny we Wroclawiu
Locations (1):
- Centrum Chorób Serca - Klinika Kardiologii, 4. Wojskowy Szpital Kliniczny, Wroclaw, Poland